CLINICAL TRIAL: NCT04420715
Title: 3D Printed Silicone Coronary Artery Simulator for Percutaneous Coronary Interventional Training
Acronym: 3DforPCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Shubin_Qiao, Director,Head of cardiology department, Fu Wai Hospital, Beijing, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018YFB1107102
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Percutaneous Coronary Intervention
Keywords: percutaneous coronary intervention; 3D printing; silicone; coronary artery simulator; training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Less-experienced group (Experimental): The participant who has completed the number of PCI less than 200 before recruiting
  Interventions: Other: Training on coronary angiography using 3D coronary artery simulator
- Experienced group (Experimental): The participant who has completed the number of PCI more than 200 before recruiting
  Interventions: Other: Training on coronary angiography using 3D coronary artery simulator

INTERVENTIONS:
Other: Training on coronary angiography using 3D coronary artery simulator — Participants will have a test of coronary arteriography before and after training, compare the scores to analysis if the simulator training is effective.

SUMMARY:
This study is aim to evaluate the feasibility and effectiveness of 3D printed silicone coronary artery simulator for percutaneous coronary interventional training.

DETAILED DESCRIPTION:
With the aging of the population, the incidence of cardiovascular diseases has exceeded that of respiratory diseases and cancer, corresponding to the rapid increase in the number of coronary stent implantation. Therefore, the standardized training of interventional cardiologists is particularly important. Nowadays percutaneous coronary intervention (PCI) training mode is mainly for the trainees to operate on the patients under the experienced operator. Although this kind of training method can truly show the operation process, it has obvious limitations. For beginners, it takes repeated training and revision to achieve proficiency and accuracy.Learning only through real surgery may result in longer operative times, increased radiation exposure, and increased complications.This study is aim to evaluate the feasibility and effectiveness of 3D printed silicone coronary artery simulator for percutaneous coronary interventional training.

ELIGIBILITY:
Inclusion Criteria:

* Previous experience in coronary intervention
* Understand the process of trail and be willing to participate

Exclusion Criteria:

* No previous experience with coronary intervention
* Unwilling to participate the trail
* Unable to complete the trail due to other problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-07 (Estimated); Primary Completion 2020-06-07 (Estimated); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
Change of the time taken in operation | Through study completion, an average of 4 hours
  The change of time taken to complete the coronary angiography assessment before and after training
Change of the amount of contrast agent used | Through study completion, an average of 4 hours
  The change of the amount of contrast agent used in the coronary angiography assessment before and after training
Change in assessment scores | Through study completion, an average of 4 hours
  The change of scores of "Rating scale of coronary angiography operation assessment" before and after training. The assessment includes operation integrity, standardization, proficiency, accuracy,etc. Every point contain 5 different levels from the worst(1) to the best(5).

CONTACTS AND LOCATIONS:
Overall Officials: Shubin Qiao, MD,PhD, Principal Investigator — Fuwai Hospital, Beijing, China
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
including the simulator details; the basic information of all participants; the scores of all participants before and after training; the training process
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after the trail completed